CLINICAL TRIAL: NCT03237286
Title: Testing a Synergistic, Neuroplasticity-Based Intervention for Depressive Neurocognition
Brief Title: Intravenous Ketamine Plus Neurocognitive Training for Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rebecca Price (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Rebecca Price, Assistant Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19040414; 1R01MH113857 (NIH)
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Depression
Keywords: depression; ketamine; neurocognitive; fMRI; cognitive training
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ketamine + Cognitive Training (Experimental)
  Interventions: Drug: Intravenous ketamine; Behavioral: Computer-based Cognitive Training
- Ketamine + Sham Training (Sham Comparator)
  Interventions: Drug: Intravenous ketamine
- Saline + Cognitive Training (Placebo Comparator)
  Interventions: Behavioral: Computer-based Cognitive Training

INTERVENTIONS:
Drug: Intravenous ketamine — Intravenous ketamine is given at a subanesthetic dose, which previous research suggests is safe and efficacious for rapid relief from depression.
  Arms: Ketamine + Cognitive Training; Ketamine + Sham Training
Behavioral: Computer-based Cognitive Training — Computer-based Cognitive Training will be delivered following intravenous ketamine to test whether learning during a post-ketamine "window of opportunity" might extend relief from depression.
  Arms: Ketamine + Cognitive Training; Saline + Cognitive Training

SUMMARY:
This study has two aims: 1) to characterize the effects of intravenous ketamine on neurocognitive markers in depressed patients; 2) to test the efficacy of a synergistic intervention for depression combining intravenous ketamine with neurocognitive training. Three of the primary outcomes listed (fMRI functional connectivity; Implicit Association Test; cognitive flexibility testing) pertain to Aim 1. For Aim 2, one primary clinical outcome (MADRS, a clinician-administered measure of depression severity) pertains to the acute (30-day) phase, while the QIDS (a self-report measure of depression severity) becomes the primary clinical outcome during the 12-month naturalistic follow-up.

DETAILED DESCRIPTION:
This study measures clinical and mechanistic outcome trajectories following ketamine (with or without adjunctive neurocognitive training) measured over an acute (30-day) period; and subsequently (for a subset of measures) over a 12-month naturalistic follow-up period.

NOTE: Corrections have been made to the "Time Frame" entries for all primary/secondary outcomes after identifying errors stemming from the study team's misunderstanding of the "Time Frame" query. Initially, the "Time Frame" query was misinterpreted to mean the range (minimum to maximum) length of the time interval over which any given assessment visit might query symptoms, and were therefore assigned erroneous values ("1 day to 2 weeks"; "1 day to lifetime") reflecting the time interval(s) queried by the instrument (e.g. at the +24 hours timepoint, symptoms are queried over a 1-day interval; at other assessment points, they could be queried over a 2-week interval for some measures, or over the entire lifetime for other measures). After recognizing this misinterpretation, the values have been adjusted to accurately reflect the a priori analytic plan.

ELIGIBILITY:
Inclusion Criteria:

Participants will:

1. be between the ages of 18 and 60 years,
2. have not responded to one or more adequate trials of FDA-approved antidepressants within the current depressive episode, determined by Antidepressant Treatment History Form
3. score ≥ 25 on the Montgomery Asberg Depression Rating Scale (MADRS)
4. score >1SD above the normative mean on the Cognitive Triad Inventory "self" subscale *OR* <1SD below the normative mean on the Rosenberg self-esteem scale
5. possess a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document
6. agree to sign a release of information (ROI), identifying another individual [friend, family member, etc.] as a contact person while the patient is enrolled in the study.

Exclusion Criteria:

1. Presence of lifetime bipolar, psychotic, or autism spectrum; current problematic substance use (e.g., substance use disorder); or lifetime recreational ketamine or PCP use
2. Use of a Monoamine Oxidase Inhibitor (MAOI) within the previous 2 weeks
3. Failure to meet standard MRI inclusion criteria: those who have cardiac pacemakers, neural pacemakers, cochlear implants, metal braces, or other non-MRI-compatible metal objects in their body, especially in the eye. Dental fillings do not present a problem. Plastic or removable dental appliances do not require exclusion. History of significant injury or surgery to the brain or spinal cord that would impair interpretation of results.
4. Current pregnancy or breastfeeding, or failure to engage in an effective birth control strategy throughout the duration of the study
5. Acute suicidality or other psychiatric crises requiring treatment escalation.
6. Changes made to treatment regimen within 4 weeks of baseline assessment
7. Reading level <6th grade
8. For study entry, patients must be reasonable medical candidates for ketamine infusion, as determined by a board-certified physician co-investigator during study screening. Serious, unstable medical illnesses including respiratory [obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics], cardiovascular [including ischemic heart disease and uncontrolled hypertension], and neurologic [including history of severe head injury] will be exclusions.
9. Clinically significant abnormal findings of laboratory parameters [including urine toxicology screen for drugs of abuse], physical examination, or ECG.
10. Uncontrolled or poorly controlled hypertension, as determined by a board-certified physician co-investigator's review of vitals collected during screening and any other relevant medical history/records.
11. Patients with one or more seizures without a clear and resolved etiology.
12. Patients starting hormonal treatment (e.g., estrogen) in the 3 months prior to Screening. Birth control is not an exclusion.
13. Past intolerance or hypersensitivity to ketamine or midazolam.
14. Patients taking medications with known activity at the NMDA or AMPA glutamate receptor [e.g., riluzole, amantadine, lamotrigine, memantine, topiramate, dextromethorphan, D-cycloserine], or the muopioid receptor.
15. Patients taking any of the following medications: St John's Wort, theophylline, tramadol, metrizamide
16. Patients who have received ECT in the past 6 months prior to Screening.
17. Patients currently receiving treatment with vagus nerve stimulation (VNS) or repetitive transcranial stimulation (rTMS).
18. Patients taking benzodiazepines (within 8 hours of infusion) or GABA agonists

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will comply with all NIMH guidelines regarding data repository/sharing.
Time Frame: We will comply with all NIMH guidelines regarding data repository/sharing.

REFERENCES:
- [Derived] Hossein S, Woody ML, Panny B, Spotts C, Wallace ML, Mathew SJ, Howland RH, Price RB. Functional connectivity subtypes during a positive mood induction: Predicting clinical response in a randomized controlled trial of ketamine for treatment-resistant depression. J Psychopathol Clin Sci. 2025 Apr;134(3):228-238. doi: 10.1037/abn0000951. Epub 2024 Sep 23. PMID 39311825
- [Derived] Price RB, Wallace ML, Mathew SJ, Howland RH. One-Year Outcomes Following Intravenous Ketamine Plus Digital Training Among Patients with Treatment-Resistant Depression: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2312434. doi: 10.1001/jamanetworkopen.2023.12434. PMID 37155171
- [Derived] Price RB, Panny B, Degutis M, Griffo A. Repeated measurement of implicit self-associations in clinical depression: Psychometric, neural, and computational properties. J Abnorm Psychol. 2021 Feb;130(2):152-165. doi: 10.1037/abn0000651. Epub 2020 Dec 3. PMID 33271040

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Started | 53 | 50 | 51
Completed | 52 | 50 | 48
Not Completed | 1 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Study withdrew participant due to repeated non-compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training | Total
Number analyzed (Participants) | 53 | 50 | 51 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.70 (10.10) | 34.60 (11.60) | 33.50 (9.90) | 34.26 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 33 | 97
  Male | 21 | 18 | 18 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 4 | 11
  Not Hispanic or Latino | 45 | 45 | 47 | 137
  Unknown or Not Reported | 3 | 3 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 2 | 7
  White | 44 | 40 | 41 | 125
  More than one race | 2 | 5 | 4 | 11
  Unknown or Not Reported | 0 | 1 | 1 | 2
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — depression severity; range 0-60; high score=worse outcome
  units on a scale | 32.28 (5.70) | 33.48 (4.90) | 32.61 (5.10) | 32.78 (5.30)
Number of failed antidepressant trials [Mean (Standard Deviation); unit: trials] — Number of adequate trials of an FDA-approved antidepressant in the current depressive episode, per Antidepressant Treatment History Form
  trials | 2.66 (1.59) | 2.60 (1.67) | 2.67 (2.46) | 2.64 (1.93)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: Trajectories from 24 hours through Day 30 post-infusion, Day 30 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 53 | 50 | 51
score on a scale | 19.72 (10.20) | 22.87 (11.63) | 23.51 (9.66)
Statistical Analysis 1: Comparison: Ketamine + Cognitive Training vs Saline + Cognitive Training; Test type: Superiority; p = .0004, Regression, Linear

2. Primary Outcome: Executive-salience Network Functional Connectivity
Description: fMRI measure (beta weights where larger beta weight = stronger connectivity)
Time Frame: Trajectories from 24 hours through Day 30 post-infusion, 24 hours reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 53 | 49 | 47
beta weights | 0.55 (0.11) | 0.59 (0.11) | 0.57 (0.10)

3. Primary Outcome: Implicit Self-representations
Description: Implicit Association Test composite difference score (performance-based measure; range = -inf-inf; high score=worse outcome; negatively signed value indicates associating oneself more strongly with positive than negative attributes)
Time Frame: Trajectories from 24 hours through Day 30 post-infusion, Day 5 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: factor score
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 51 | 43 | 44
factor score | -.16 (1.00) | 0.15 (1.03) | 0.03 (0.97)

4. Primary Outcome: Cognitive Flexibility
Description: Neurocognitive testing via NIH Toolbox DCCS fully-corrected T-scores (range = 0-100; high score=better outcome)
Time Frame: Trajectories from 24 hours through Day 30 post-infusion, Day 30 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 37 | 35 | 36
score on a scale | 54.51 (13.33) | 49.34 (12.48) | 53.25 (12.98)

5. Primary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: Trajectories from Day 30 through 12 months post-infusion (naturalistic follow-up), Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 26 | 29 | 26
score on a scale | 10.77 (6.84) | 12.03 (5.94) | 10.42 (4.38)

6. Secondary Outcome: Executive-salience Network Functional Connectivity During Resting State
Description: fMRI measure (beta weights where larger beta weight = stronger connectivity)
Time Frame: Trajectories from 24 hours through Day 30 post-infusion, 24 hours reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 53 | 49 | 47
beta weights | 0.53 (0.10) | 0.50 (0.09) | 0.51 (0.12)

7. Secondary Outcome: Affective Flexibility
Description: 'D-Prime' discrimination Z-score measured via accuracy of responses during the Affective Go/No-Go task (range: -inf-inf; high score=better performance; Z-score of 0=the sample mean)
Time Frame: Trajectories from 24 hours through Day 30 post-infusion, Day 30 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 45 | 43 | 43
Z-score | -.18 (1.71) | -.07 (1.52) | 0.26 (1.62)

8. Secondary Outcome: PROMIS Measures-depression
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported depression T-score range: 0-100 (higher score = worse outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 35 | 38 | 35
score on a scale | 58.97 (12.15) | 61.01 (9.54) | 57.13 (9.57)

9. Secondary Outcome: PROMIS Measures-anxiety
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported anxiety T-score range: 0-100 (higher score = worse outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 35 | 38 | 35
score on a scale | 58.07 (9.42) | 62.49 (9.26) | 57.88 (8.87)

10. Secondary Outcome: PROMIS Measures-anger
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported anger T-score range: 0-100 (higher score = worse outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 35 | 38 | 35
score on a scale | 50.27 (13.03) | 54.21 (10.44) | 49.59 (10.23)

11. Secondary Outcome: PROMIS Measures-positive Affect
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported positive affect/well-being T-score range: 0-100 (higher score = better outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 35 | 38 | 35
score on a scale | 44.12 (7.72) | 44.02 (7.76) | 45.98 (7.60)

12. Secondary Outcome: PROMIS Measures-sleep Disturbance
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported sleep disturbance T-score range: 0-100 (higher score = worse outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 35 | 38 | 35
score on a scale | 53.06 (9.91) | 53.78 (8.63) | 51.41 (10.29)

13. Secondary Outcome: PROMIS Measures-cognitive Function
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported cognitive function T-score range: 0-100 (higher score = better outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 36 | 38 | 35
score on a scale | 43.61 (9.54) | 39.19 (8.07) | 44.87 (8.81)

14. Secondary Outcome: PROMIS Measures-substance Use
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported substance use Raw score range: 0-35 (higher score = worse outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 34 | 38 | 35
score on a scale | 3.00 (5.22) | 2.32 (5.09) | 3.03 (5.94)

15. Secondary Outcome: PROMIS Measures-alcohol
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported alcohol use T-score range: 0-100 (higher score = worse outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 35 | 38 | 35
score on a scale | 46.29 (8.56) | 47.82 (5.35) | 47.25 (7.04)

16. Secondary Outcome: Cognitive Triad Inventory
Description: Negative perceptions of self, future, & world (range=36-252; higher score = better outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 36 | 38 | 35
score on a scale | 133.89 (35.15) | 126.00 (39.02) | 138.97 (28.50)

17. Secondary Outcome: Columbia-Suicide Severity Rating Scale
Description: Suicidality and patient safety (most severe ideation score, range=0-5; higher score = worse outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 27 | 30 | 29
score on a scale | 0.70 (1.14) | 1.30 (1.24) | 1.10 (1.29)

18. Secondary Outcome: WHO Disability Assessment Scale (SR)
Description: Global functioning (range=0-48; higher score = worse outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 33 | 36 | 33
score on a scale | 10.58 (9.28) | 15.75 (10.87) | 12.64 (10.72)

19. Secondary Outcome: Cognitive Flexibility Scale
Description: Self-reported cognitive flexibility (range=12-72; higher score = better outcome)
Time Frame: Trajectories from 24 hours through Month 12 post-infusion, Month 12 reported
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Saline + Cognitive Training
Number analyzed (Participants) | 36 | 38 | 35
score on a scale | 52.64 (8.82) | 50.82 (10.81) | 51.20 (10.46)

20. Secondary Outcome: Neuroplasticity-related Markers in Blood
Description: ketamine metabolite (2R,6R)-HNK concentration levels (range=0-inf; higher score = greater concentration in blood)
Time Frame: 40min post-infusion
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 50 | 50
ng/mL | 26.94 (11.59) | 27.35 (11.76)

ADVERSE EVENTS:
Time Frame: 4 hours
Description: Adverse events collected using the Patient Rated Inventory of Side Effects (PRISE; Rush et al 2004) supplemented by open-ended questions. AEs were tallied for new or worsening symptoms (relative to pre-infusion baseline) with onset on the infusion day. Tallies are combined across two arms (ketamine+sham, ketamine+cognitive training) because the collected AEs pertain specifically to the drug infusion; the cognitive or sham behavioral training did not begin until AFTER AEs were reported/collected.
Groups:
- Ketamine: Includes all participants receiving the study drug (0.5 mg/kg IV ketamine over 40min), irrespective of Cognitive Training condition (active and sham collapsed)
- Saline: Includes all participants receiving a placebo infusion of saline (over 40min). All participants in this arm later went on to receive the active Cognitive Training condition.
Arm/Group | Ketamine | Saline
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/51
Other Adverse Events (participants affected / at risk) | 102/103 | 38/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=103) | Saline (N=51)
anxiety (Psychiatric disorders) | 10 | 2
decreased energy (General disorders) | 16 | 3
difficulty focusing vision (Nervous system disorders) | 2 | 0
difficulty sleeping: too little (Psychiatric disorders) | 1 | 1
difficulty sleeping: too much (Psychiatric disorders) | 5 | 4
difficulty urinating (Renal and urinary disorders) | 1 | 0
dissociative effects (Psychiatric disorders) | 100 | 11
dizziness (Nervous system disorders) | 70 | 10
dry mouth (Gastrointestinal disorders) | 40 | 5
elevated blood pressure (Cardiac disorders) | 7 | 2
elevated heart rate (Cardiac disorders) | 3 | 0
emesis (Gastrointestinal disorders) | 4 | 0
emotional indifference (Psychiatric disorders) | 8 | 1
feeling "discombobulated" (General disorders) | 1 | 0
feeling "high" (per verbal report) (Psychiatric disorders) | 1 | 0
headache (Nervous system disorders) | 17 | 4
increased appetite (Gastrointestinal disorders) | 12 | 1
increased weight (Metabolism and nutrition disorders) | 1 | 0
loss of sexual desire (Reproductive system and breast disorders) | 2 | 0
lowered pulse (Cardiac disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 31 | 7
palpitations (Cardiac disorders) | 11 | 0
restlessness (General disorders) | 18 | 2
suicidal ideation (Psychiatric disorders) | 1 | 0
sweating (General disorders) | 18 | 3
tinnitus (Nervous system disorders) | 1 | 0
tremors (Nervous system disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT03237286/Prot_SAP_000.pdf